CLINICAL TRIAL: NCT05223179
Title: Randomised, Double-blind, Placebo-controlled, Dose-escalation Study of the Safety, Tolerability, and Immunogenicity of Intramuscular CodaVax-H1N1 in Healthy Adults
Brief Title: Intramuscular CodaVax-H1N1 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CDX-FLU-103
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Influenza, Human
Keywords: Influenza, Human; Viral Vaccines; Vaccines, Live Attenuated
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CODA-VAX H1N1 (Experimental): Live Attenuated Vaccine administered by Intramuscular Injection
  Interventions: Biological: CODA-VAX H1N1
- Flucelvax Quad (Active Comparator): Licensed Injectable Seasonal Influenza Vaccine
  Interventions: Biological: Flucelvax Quad
- Saline (Placebo Comparator): Normal Sterile Saline for Intramuscular Injection
  Interventions: Other: Saline

INTERVENTIONS:
Biological: CODA-VAX H1N1 — Intramuscular Live Attenuated Influenza H1N1 Vaccine
  Arms: CODA-VAX H1N1
Biological: Flucelvax Quad — Licensed Seasonal Injectable Influenza Vaccine
  Arms: Flucelvax Quad
Other: Saline — Saline
  Arms: Saline

SUMMARY:
This study is a Phase 1, 2-part, randomised, double-blind, controlled, clinical trial to evaluate the safety and immune response of CodaVax-H1N1 in healthy adults aged 18 to 49 years. Participants will be enrolled in autumn 2022 (southern hemisphere) and followed through the 2022 influenza season (Part A) or enrolled in autumn 2023 and followed through the 2023 influenza season (Part B). Participants will be screened within 28 days of randomization, and eligible participants in Part A will be enrolled into 1 of 3 sequential cohorts and randomised to receive a single dose of CodaVax-H1N1, placebo (normal saline), or licenced injectable seasonal influenza vaccine (Flucelvax Quad). Each subsequent cohort will include a higher dose of CodaVax H1N1 than the previous cohort, in addition to placebo and the licensed injectable seasonal influenza vaccine. In Part B, 24 eligible participants will be enrolled into 1 of 2 sequential cohorts and randomised to receive a single IM dose of CodaVax-H1N1 or placebo.

DETAILED DESCRIPTION:
This study is a Phase 1, 2-part, randomised, double-blind, controlled, clinical trial to evaluate the safety and immune response of CodaVax-H1N1 in healthy adults aged 18 to 49 years. Participants will be enrolled in autumn 2022 (southern hemisphere) and followed through the 2022 influenza season (Part A) or enrolled in autumn 2023 and followed through the 2023 influenza season. Participants will be screened within 28 days of randomization, and eligible participants in Part A will be enrolled into 1 of 3 sequential cohorts and randomised to receive a single dose of CodaVax-H1N1, placebo (normal saline), or licensed injectable seasonal influenza vaccine (Flucelvax Quad). Each subsequent cohort will include a higher dose of CodaVax H1N1 than the previous cohort, in addition to placebo and the licensed injectable seasonal influenza vaccine. In Part B, 24 eligible participants will be enrolled into 1 of 2 additional sequential cohorts and randomised to receive a single IM dose of CodaVax-H1N1 or placebo.

Participants will record reactogenicity events (local events, systemic events, and temperature) in a daily diary for 7 days after the dose. Each participant will be contacted by telephone on the day after dosing for safety assessment and review of the diary data. Participants will return to the clinic on Days 4, 8, 29, 91, and 181 for safety and immune response assessments.

All adverse events and concomitant medications will be recorded from signing of the informed consent form (ICF) to 28 days postdose. After 28 days until the end of the study, only medically attended adverse events (MAAEs), new onset chronic illnesses (NCIs), serious adverse events (SAEs), immunosuppressive medications, blood products like transfusions or infusions, and vaccines will be recorded. A complete physical examination will be performed at Screening, and targeted and symptom-driven physical examinations will be performed predose on Day 1, 2 hours postdose, and at each postdose visit through Day 91. Vital signs will be measured at the same time points. An electrocardiogram (ECG) will be performed at Screening and on Day 29.

A serum sample will be collected predose and on Days 29, 91, and 181 for measurement of immune response.

A whole blood sample will be collected predose and on Day 8 and PBMCs isolated for measurement of T-cell response.

If a participant experiences acute symptoms compatible with viral respiratory infection, nasopharyngeal swab samples will be collected for a rapid influenza diagnostic test and respiratory virus PCR assay panel (including SARS-CoV-2) as indicated for symptomatic respiratory infection and will perform the rapid influenza diagnostic test.

The primary analysis of study data will be conducted after all participants complete the Day 29 visit. The final analysis will be conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18 and ≤ 35 kg/m2
* In good health with no history, or current evidence, of clinically significant medical conditions
* Negative SARS-CoV-2 test predose on Day 1
* For all women, negative pregnancy test
* Agreement to comply with conditions to prevent the spread of genetically modified organisms (GMOs)

Exclusion Criteria:

* Pregnant or lactating women or women who plan to become pregnant through Day 29
* Inadequate venous access for repeated phlebotomy
* History of severe reaction to vaccination
* Receipt of any licenced or investigational influenza vaccine within 6 months before Day 1
* Receipt of any live vaccine within 30 days before Day 1
* Tattoo, skin reaction, or other condition at the injection site that would interfere with assessment of local reactogenicity

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability by Assessing Percentage of Participants with Reactogenicity Events | Reactogenicity events from Day 1 to Day 7
  Percentage of participants with reactogenicity events
Safety and Tolerability by Assessing Percentage of Participants with Adverse Events | Adverse events (AEs) from Day 1 to Day 29
  Percentage of participants with adverse events
Safety and Tolerability by Assessing Percentage of Participants with MAAEs, NCIs, and SAEs. | MAAEs, NCIs, SAEs from Day 1 to Day 181
  Percentage of participants with MAAEs, NCIs, and SAEs.

SECONDARY OUTCOMES:
Humoral Immunogenicity | HAI assay titre against A/California/07/2009 and the current seasonal influenza vaccine H1N1 and H3N2 strains measured in samples collected on Days 1, 29, 91, and 181
  To assess the humoral immunogenicity elicited by CodaVax-H1N1 at nominal doses of 5×104, 5×105, and 5×106 PFU by IM injection

CONTACTS AND LOCATIONS:
Locations (1):
- Lis Gilmour, Senior Project Manager, Morayfield, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No